CLINICAL TRIAL: NCT00935623
Title: Development of a Safe and Reproducible Human Sporozoite Challenge Model for Plasmodium Vivax in Healthy Adults in the United States
Brief Title: Clinical Trial for the Development of a Safe Malaria Challenge Model That Can be Reproduced in Humans
Acronym: Pvivax
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: United States Department of Defense (U.S. Federal Agency); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: WRAIR 1518; HSRRB A-15209 (Other: USAMRMC)
Record Dates: First submitted 2009-07-07; First posted 2009-07-09 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Plasmodium Vivax Malaria
Keywords: Malaria, Plasmodium vivax
MeSH Terms: conditions — Malaria, Vivax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): The first cohort will be challenged with 5 bites from P. vivax-infected mosquitoes each carrying at least a grade 2 sporozoite infection (>10 sporozoites in salivary gland).
  Interventions: Biological: Malaria Challenge
- Cohort 2 (Experimental): If the first cohort has less than 100% infectivity rate, the second cohort will be challenged with up to 10 grade 2 infective bites to ensure 100% infectivity rate.
  Interventions: Biological: Malaria Challenge

INTERVENTIONS:
Biological: Malaria Challenge — Malaria challenge

SUMMARY:
The purpose of this study is to demonstrate that volunteers can be safely and reproducibly infected with Plasmodium vivax (P. vivax) by the bites of experimentally infected Anopheles dirus (An. dirus) mosquitoes carrying P. vivax sporozoites in their salivary glands.

DETAILED DESCRIPTION:
The study is a proof-of-concept clinical investigation designed to develop a safe and practical sporozoite challenge model for Plasmodium vivax in humans with a goal of 100% infectivity rate. The development and standardization of such a model will make possible efficacy evaluations of candidate P. vivax vaccines in Phase 2a trials. This trial is conducted in collaboration with Armed Forces Research Institute of Medical Sciences (AFRIMS) investigators in Bangkok, Thailand, who will be recruiting adult blood donors from a pool of patients who present with active P. vivax infections in Thailand. Samples of P. vivax infected blood will be collected and fed via membrane feeding apparatus to colony-reared Anopheles dirus mosquitoes at the AFRIMS Entomology Lab. A portion of the same blood will meanwhile be screened for potential co-infections at the AFRIMS Retrovirology Laboratory. When screening tests have confirmed the presence of only P. vivax in the blood (no co-infections with other malaria species), and selected dissection on days 3-7 has revealed oocyst production in the blood-fed mosquitoes, the mosquitoes will be transported from the AFRIMS insectary in Thailand to the WRAIR insectary in the US by a standard procedure (herein described) including permits and assurance against accidental release of the infected mosquitoes. Transport will be conducted in compliance with Thai exporting and US importing requirements.

Our study will involve two cohorts, each to be challenged once, in the hope of demonstrating reproducibility of the entire challenge procedure. Each cohort comprises up to 6 healthy adult volunteers. The first cohort will be challenged with 5 bites from P. vivax-infected mosquitoes each carrying at least a grade 2 sporozoite infection (>10 sporozoites in salivary gland).

If all six volunteers in the first cohort develop P. vivax infection, the same procedure will be repeated in the second cohort. If the first cohort has less than 100% infectivity rate, the second cohort will be challenged with up to 10 grade 2 infective bites to ensure 100% infectivity rate. Volunteers will be closely monitored post-infection, and will be treated with standard chloroquine and primaquine therapies when the infection becomes patent in the peripheral blood.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults (male or non-pregnant, non-lactating female) 18 to 55 years of age;
* Able to provide free and willing written informed consent to participate;
* A score at least 80% correct on a 10 question Assessment of Understanding;
* No plans to travel to a malaria endemic area during the course of the study;
* Duffy positive phenotype;
* Normal (non-deficient) G6PD phenotype (range : 4.6 to 13.5 u/gm hemoglobin);
* Free of significant health problems as established by medical history and clinical examination completed prior to the study;
* Available to participate and reachable by phone for duration of study (approximately 9 months starting from screening).
* Only subjects with no or low cardiac risk factors according to the Gaziano study and a normal EKG will be included in the study

Exclusion Criteria:

* Pregnant or nursing at screening or plans to become pregnant or nurse from the time of enrollment until 6 months after sporozoite challenge;
* Duffy negative phenotype;
* G6PD deficiency or have any hemoglobinopathy by history;
* Past infection with any species of malaria (as demonstrated by a positive thick smear) in the last 5 years;
* History of receipt of treatment or prophylaxis for malaria during the previous 6 months;
* History of receipt of malaria vaccine within the previous 5 years;
* History of receipt of malaria challenge (being bitten by experimentally infected mosquitoes) within the previous 5 years;
* Plans to travel to malarious areas during the study period;
* Allergy to antimalarials or significant (e.g. systemic) hypersensitivity reactions to mosquito bites (local hypersensitivity reactions at the site of a mosquito bite are not an exclusion criterion);
* History of psoriasis (given its interaction with chloroquine);
* Use of any investigational or non-registered drug or vaccine within 30 days preceding the challenge or planned use during the study period;
* Use or planned use of any drugs with significant anti-malarial activity, such as doxycycline, clindamycin, azithromycin, during the study period (volunteers can withhold the use of these medications during the study period, at the minimum starting from 4 weeks before the challenge until 4 weeks after becoming parasitemic);
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including HIV infection and history of splenectomy;
* Administration of chronic (defined as more than 14 days) immunosuppressants or other immune-modifying drugs within six months of challenge;

  * For corticosteroids, this is defined as prednisone, or equivalent, 0.5 mg/kg/day;
  * Inhaled and topical steroids are allowed;
* A family history of congenital or hereditary immunodeficiency;
* Chronic or active neurologic disease including seizure disorder;
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic, or renal functional abnormality, as determined by medical history, physical examination, or abnormal baseline laboratory screening tests:

  * ALT above normal range (table 9);
  * Creatinine above normal range (table 9);
  * Hemoglobin below normal range (table 10);
  * Platelet count below normal range (table 10);
  * Total white cell count below normal range (table 10);
* Acute disease at the time of enrollment

  * Acute disease is defined as the presence of a moderate or severe illness with or without fever;
  * Challenge can be administered to persons with a minor illness, such as diarrhea or mild upper respiratory infection without fever (i.e., oral temperature < 38°C/100.4°F);
* Hepatomegaly, right upper quadrant abdominal pain or tenderness;
* Seropositive for HIV, hepatitis C virus (antibodies to HIV and HCV), and/or HBsAg;
* Administration of immunoglobulins and/or any blood products within the 3 months preceding challenge or planned administration during the study period;
* Suspected or known current alcohol abuse/drug abuse as obtained by history and physical examination;
* Inability to make follow-up visits;
* Any other significant finding that in the opinion of the investigator would increase the risk of having an adverse outcome from participating in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-04-21 (Actual); Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Detection of erythrocytic stage P. vivax parasites by blood smear in volunteers during the 28 day period post challenge via the bites of five P. vivax-infected mosquitoes; Occurrence and intensity of solicited and unsolicited symptoms post challenge | 28 days post challenge

SECONDARY OUTCOMES:
Parasitologic and clinical infections in challenge volunteers will be characterized by descriptive analysis of prepatent and patent periods, incubation period and time to resolution of signs and symptoms, and timing and number of relapses. | Cross-sectional

CONTACTS AND LOCATIONS:
Overall Officials: Ilin Chuang, MD, MPH, Principal Investigator — US Military Malaria Vaccine Program, Naval Medical Research Center
Locations (1):
- WRAIR Clinical Trials Center, Silver Spring, Maryland, United States